CLINICAL TRIAL: NCT07180563
Title: Randomized Controlled Trial of Berberine in Combination With Doxycycline in the Treatment of Chronic Endometritis
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY-2024-246
Record Dates: First submitted 2025-03-20; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-03

CONDITIONS: Chronic Endometritis
MeSH Terms: interventions — Doxycycline

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- At present, the commonly used clinical treatment for chronic endometritis is oral doxycycline (Active Comparator): At present, the commonly used clinical treatment for chronic endometritis is oral doxycycline
  Interventions: Drug: At present, the commonly used clinical treatment for chronic endometritis is oral doxycycline
- Participants were treated with doxycycline + berberin for chronic endometritis (intervention group) (Experimental): Participants were treated with doxycycline + berberin for chronic endometritis (intervention group)
  Interventions: Drug: Participants were treated with doxycycline + berberin for chronic endometritis (intervention group).

INTERVENTIONS:
Drug: Participants were treated with doxycycline + berberin for chronic endometritis (intervention group). — Diagnosed chronic endometritis according to endometrial biopsy pathology , the specific medication plan for the intervention group was to use doxycycline 100mg, bid + berberin 100mg, tid, continuously for 14 days.
  Arms: Participants were treated with doxycycline + berberin for chronic endometritis (intervention group)
Drug: At present, the commonly used clinical treatment for chronic endometritis is oral doxycycline — 11After hysteroscopic diagnosis of chronic endometritis, patients received monotherapy with doxycycline hydrochloride capsules for 14 days.
  Arms: At present, the commonly used clinical treatment for chronic endometritis is oral doxycycline

SUMMARY:
Study Subjects: Eligible patients were initially diagnosed with chronic endometritis (CE) by CD138 testing through outpatient hysteroscopy. Positive CD138 expression is defined as at least one or more positive-staining plasma cells per 10 high-power fields identified as positive, and less than one positive-stained plasma cell identified as negative [8]. All patients signed an informed consent form prior to participating in the study, and the study followed the principles of the Declaration of Helsinki.

Inclusion Criteria: Diagnosis of chronic endometritis by CD138 immunohistochemistry; Age≥ 20 years old, females of childbearing age; Agree to undergo hysteroscopy and hysteroscopic endometrial biopsy; No serious systemic disease; There are no contraindications to oral administration of doxycycline hydrochloride and berberine hydrochloride.

Exclusion criteria: patients with pregnancy status, uterine malignant disease, hormone therapy within 3 months, glucose-6 phosphate dehydrogenase deficiency, hemolytic anemia, hypersensitivity to berberine hydrochloride or doxycycline. In addition, berberine hydrochloride has fewer oral adverse reactions, occasional nausea and vomiting, rash and drug fever, which disappear after stopping the drug. If the patient takes the wrong or missed medication, it is excluded.

Withdrawal criteria: If the patient has corresponding adverse reaction symptoms, those with mild symptoms can be temporarily observed, and if the symptoms are severe, they can be transferred to the Department of Gastroenterology for diagnosis and treatment, and those who need to stop the drug will be withdrawn from this study.

DETAILED DESCRIPTION:
Grouping: The patients were randomly divided into the experimental group and the control group by a simple numerical table method, with a ratio of 1:1.

* Patients in the experimental group were treated with berberine hydrochloride tablets (0.1g*100 tablets/bottle, Shenyang First Pharmaceutical Co., Ltd., Northeast Pharmaceutical Group) + doxycycline hydrochloride capsules (100mg*24 tablets/box, Guangzhou Percello Pharmaceutical Co., Ltd.), with oral administration of berberine hydrochloride tablets 100mg Tid per day and oral administration of doxycycline hydrochloride capsules 100mg Bid per day for 14 days.
* Patients in the control group were treated with oral doxycycline hydrochloride capsules only and oral doxycycline hydrochloride capsules 100 mg twice a day for 14 days.

Evaluation indicators: Patients in both groups started taking antibiotics after being diagnosed with chronic endometritis by CD138 detection. After a course of treatment, the conversion rate of chronic endometritis expression from positive to negative was compared between the two groups.

Outcomes: Primary outcomes: Cure rate of chronic endometritis; Secondary outcomes: Number of CD138 positives per 10 high-power fields; Recurrence rate of uterine polyps, number and size of uterine polyps recurrence.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of chronic endometritis by CD138 immunohistochemistry; Age≥ 20 years old, females of childbearing age; Agree to undergo hysteroscopy and hysteroscopic endometrial biopsy; No serious systemic disease; There are no contraindications to oral administration of doxycycline hydrochloride and berberine hydrochloride.

Exclusion Criteria:

Patients with pregnancy status, uterine malignant disease, hormone therapy within 3 months, glucose-6 phosphate dehydrogenase deficiency, hemolytic anemia, hypersensitivity to berberine hydrochloride or doxycycline. In addition, berberine hydrochloride has fewer oral adverse reactions, occasional nausea and vomiting, rash and drug fever, which disappear after stopping the drug. If the patient takes the wrong or missed medication, it is excluded.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 206 (Estimated)
Dates: Start 2025-03-15 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Patients in both groups started taking antibiotics after being diagnosed with chronic endometritis by CD138 testing. After a course of treatment, the conversion rate of chronic endometritis expression from positive to negative was compared between the tw | One month

SECONDARY OUTCOMES:
Number of CD138 positives per 10 high-power fields; recurrence rate of uterine polyps; Number and size of recurrence of uterine polyps. | One month

CONTACTS AND LOCATIONS:
Locations (1):
- The Fourth Affiliated Hospital of Zhejiang University School of Medicine, Yiwu, Zhejiang, China

REFERENCES:
- [Result] McQueen DB, Bernardi LA, Stephenson MD. Chronic endometritis in women with recurrent early pregnancy loss and/or fetal demise. Fertil Steril. 2014 Apr;101(4):1026-30. doi: 10.1016/j.fertnstert.2013.12.031. Epub 2014 Jan 23. PMID 24462055
- [Result] Cicinelli E, Matteo M, Tinelli R, Lepera A, Alfonso R, Indraccolo U, Marrocchella S, Greco P, Resta L. Prevalence of chronic endometritis in repeated unexplained implantation failure and the IVF success rate after antibiotic therapy. Hum Reprod. 2015 Feb;30(2):323-30. doi: 10.1093/humrep/deu292. Epub 2014 Nov 10. PMID 25385744
- [Result] Hirata K, Kimura F, Nakamura A, Kitazawa J, Morimune A, Hanada T, Takebayashi A, Takashima A, Amano T, Tsuji S, Kaku S, Kushima R, Murakami T. Histological diagnostic criterion for chronic endometritis based on the clinical outcome. BMC Womens Health. 2021 Mar 4;21(1):94. doi: 10.1186/s12905-021-01239-y. PMID 33663485
- [Result] Chen YX, Gao QY, Zou TH, Wang BM, Liu SD, Sheng JQ, Ren JL, Zou XP, Liu ZJ, Song YY, Xiao B, Sun XM, Dou XT, Cao HL, Yang XN, Li N, Kang Q, Zhu W, Xu HZ, Chen HM, Cao XC, Fang JY. Berberine versus placebo for the prevention of recurrence of colorectal adenoma: a multicentre, double-blinded, randomised controlled study. Lancet Gastroenterol Hepatol. 2020 Mar;5(3):267-275. doi: 10.1016/S2468-1253(19)30409-1. Epub 2020 Jan 8. PMID 31926918
- [Result] Shakeri F, Kiani S, Rahimi G, Boskabady MH. Anti-inflammatory, antioxidant, and immunomodulatory effects of Berberis vulgaris and its constituent berberine, experimental and clinical, a review. Phytother Res. 2024 Apr;38(4):1882-1902. doi: 10.1002/ptr.8077. Epub 2024 Feb 15. PMID 38358731
- [Result] Kuroda K, Takamizawa S, Motoyama H, Tsutsumi R, Sugiyama R, Nakagawa K, Sugiyama R, Kuribayashi Y. Analysis of the therapeutic effects of hysteroscopic polypectomy with and without doxycycline treatment on chronic endometritis with endometrial polyps. Am J Reprod Immunol. 2021 Jun;85(6):e13392. doi: 10.1111/aji.13392. Epub 2021 Jan 27. PMID 33501741
- [Result] Singh N, Sethi A. Endometritis - Diagnosis,Treatment and its impact on fertility - A Scoping Review. JBRA Assist Reprod. 2022 Aug 4;26(3):538-546. doi: 10.5935/1518-0557.20220015. PMID 35621273